CLINICAL TRIAL: NCT00635037
Title: Acupuncture Versus Trigger Point Injection Combined With Dipyrone and Cyclobenzaprine on Pain Relief of Patients With Myofascial Pain: Randomized Clinical Study
Brief Title: Myofascial Pain:Acupuncture Versus Trigger Point Injection Combined With Dipyrone and Cyclobenzaprine
Acronym: ACP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Adriana Machado Issy/ Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACP myofascial; No grant
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Myofascial Pain Syndromes
Keywords: Myofascial pain syndrome; Acupuncture; Nonsteroidal anti-inflammatory agents; Muscle relaxants, central; Quality of life.; muscle relaxants, analgesia
MeSH Terms: conditions — Myofascial Pain Syndromes; Muscle Hypotonia; Agnosia | interventions — Bupivacaine; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): G1 (n=15)received trigger point injection of 0.25% bupivacaine (1 ml/point) twice a week, 10 mg/day cyclobenzaprine and 500 mg dipyrone every 8 h.
  G2(n=15) was submitted to classical and trigger point acupuncture twice a week.
  Interventions: Drug: bupivacaine and acupuncture

INTERVENTIONS:
Drug: bupivacaine and acupuncture — * trigger point injection of 0.25% bupivacaine (1 ml/point) twice a week, 10 mg/day cyclobenzaprine and 500 mg dipyrone every 8 h.
  * acupuncture twice a week

SUMMARY:
CONTEXT AND OBJECTIVE: Myofascial syndrome is the most frequent condition of chronic pain. The objective of the present study was to compare the analgesic action of acupuncture and trigger point injection combined with cyclobenzaprine and dipyrone.

DESIGN AND SETTING: A randomized study was performed at the Pain Clinic. METHODS: Thirty patients were divided into two groups: G1 received trigger point injection of 0.25% bupivacaine (1 ml/point) twice a week, 10 mg/day cyclobenzaprine and 500 mg dipyrone every 8 h. G2 was submitted to classical and trigger point acupuncture twice a week. The patients were asked to continue physical exercise. The following parameters were evaluated: pain intensity rated on a numerical and verbal scale, quality of life before and four weeks after treatment, and quality of analgesia.

DETAILED DESCRIPTION:
Among the 39 patients selected, nine (3 in group 1 and 6 in group 2) were excluded from the study because they did not attend the visits scheduled for the procedures and assessment or because they did not respond to the questionnaires.

ELIGIBILITY:
Inclusion Criteria:- patients of both genders

* chronic myofascial syndrome (duration of more than three months),
* ranging in age from 18 to 65 year,
* pain intensity score of 3 or higher (rated on a numerical scale ranging from 0 to 10)

Exclusion Criteria:

* patients with disc herniation,
* osteoarthritis,
* vertebral collapse,
* temporomandibular joint dysfunction,
* infection, -
* tumors,
* coagulopathy, -
* psychiatric disease,
* cognitive disorders.
* Patients who had used any type of analgesic or muscle relaxant agent 15 days before the study and those taking anticoagulants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2005-02 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Pain relief | 1year

SECONDARY OUTCOMES:
compare the analgesic action of acupuncture and trigger point injection combined with cyclobenzaprine and dipyrone | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Miriam CB Gazi, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Pain Setor of Federal University of Sao Paulo, São Paulo, São Paulo, Brazil